CLINICAL TRIAL: NCT02495207
Title: A Histo-immunological Comparative Study of Bone Cutting by Conventional Surgery and Piezosurgery on the Secretion of Heat Shock Protein 70 (HSP70) and on the Bone Cells
Brief Title: A Comparison Between Conventional Surgery and Piezosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDDS-OMFS-03-2015
Record Dates: First submitted 2015-06-19; First posted 2015-07-13 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Third Molars Extraction
MeSH Terms: interventions — Piezosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Surgery (No Intervention): No intervention in this arm. The patients are going to undergo normal surgical intervention. Conventional surgery will be performed to extract the impacted third molars.
- Piezosurgery (Experimental): Patients here will undergo a piezosurgery to extract their third molars on both sides.
  Interventions: Device: Piezosurgery

INTERVENTIONS:
Device: Piezosurgery — This intervention is dependent on use of piezosurgery to conduct the required bone cuts to remove third molars.
  Arms: Piezosurgery

SUMMARY:
Evaluation of the effect of conventional and piezo-surgery on the secretion of Heat Shock Protein (HSP70) and on the vial bone cells at the peripheral bone cut sides after the removal of impacted mandibular third molars on both sides of the jaw.

DETAILED DESCRIPTION:
The study is about measuring the amount of HSP70 using Elisa kit for detecting HSP70 and mason trichrome for histological findings in which the study samples are patients who have bilateral impacted mandibular third molar to be extracted with bone removal. First we collect bone sample for mason trichrome with either method then we collect the second samples after removing most of the bones cover the impacted third molar for checking HSP70 levels. Then the bone samples are treated using a special protocol to eliminate the protein from bone samples for the Elisa analysis. The other bone samples are going to be studied under the microscope.

ELIGIBILITY:
Inclusion Criteria:

* bilateral identical impacted third molar that need at least 3 mm of bone removal

Exclusion Criteria:

* Pregnancy
* Smokers
* Infectious diseases
* Infections around third molars (i.e. pericoronitis).
* Alcoholic patients

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-03-14 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Levels of Heat Shock Protein 70 | Five minutes before third molar removal with the last removed layer of bone
  This will be measured using ELISA methodology

SECONDARY OUTCOMES:
Percentage of viable bone cells | This variable will be measured from the specimens taken within the first 15 minutes of bone cutting to remove third molars
  Percentage of viable bone cells will be calculated based on the counts of viable bone cells observed under the microscope.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Al-buzem, DDS, Principal Investigator — MSc student, Oral and Maxillofacial Department, University of Damascus Dental School
Locations (1):
- Department of Oral and Maxillofacial Surgery, University of Damascus Dental School, Damascus, Damscus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sivolella S, Berengo M, Bressan E, Di Fiore A, Stellini E. Osteotomy for lower third molar germectomy: randomized prospective crossover clinical study comparing piezosurgery and conventional rotatory osteotomy. J Oral Maxillofac Surg. 2011 Jun;69(6):e15-23. doi: 10.1016/j.joms.2010.12.036. Epub 2011 Mar 21. PMID 21419542
- [Background] Mantovani E, Arduino PG, Schierano G, Ferrero L, Gallesio G, Mozzati M, Russo A, Scully C, Carossa S. A split-mouth randomized clinical trial to evaluate the performance of piezosurgery compared with traditional technique in lower wisdom tooth removal. J Oral Maxillofac Surg. 2014 Oct;72(10):1890-7. doi: 10.1016/j.joms.2014.05.002. Epub 2014 May 13. PMID 25234524
- [Background] Rullo R, Addabbo F, Papaccio G, D'Aquino R, Festa VM. Piezoelectric device vs. conventional rotative instruments in impacted third molar surgery: relationships between surgical difficulty and postoperative pain with histological evaluations. J Craniomaxillofac Surg. 2013 Mar;41(2):e33-8. doi: 10.1016/j.jcms.2012.07.007. Epub 2012 Aug 11. PMID 22890087
- [Background] Gulnahar Y, Huseyin Kosger H, Tutar Y. A comparison of piezosurgery and conventional surgery by heat shock protein 70 expression. Int J Oral Maxillofac Surg. 2013 Apr;42(4):508-10. doi: 10.1016/j.ijom.2012.10.027. Epub 2012 Nov 26. PMID 23196065
- [Background] Gulnahar Y, Kosger HH, Tutar Y. The role of preoperative oxidative stress and mandibular third molar postoperative outcome--reply. Int J Oral Maxillofac Surg. 2013 Nov;42(11):1500-1. doi: 10.1016/j.ijom.2013.07.002. Epub 2013 Aug 1. No abstract available. PMID 23916119